CLINICAL TRIAL: NCT06676514
Title: Evaluation of the Efficacy of Clostridium Butyricum CBM588® on Symptoms and Quality of Life in Patients With Diarrhea-dominant Irritable Bowel Syndrome (PROREDI: (PRObiotic REmedy for DIarrhea)
Brief Title: Study to Evaluate the Treatment Benefits of Probiotic Clostridium Butyricum CBM588® for IBS-D
Acronym: PROREDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104_7maggio2023_Clostrydium
Record Dates: First submitted 2024-11-02; First posted 2024-11-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: IBS-D (Diarrhea-predominant)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): This group received probiotic treatment for IBS-D as three tablets daily for 8-weeks
  Interventions: Dietary Supplement: Probiotic Clostridium butyricum CBM588®
- Control group (Active Comparator): This group received standard of care treatment for IBS-D.
  Interventions: Other: Standard of care IBS-D treatment

INTERVENTIONS:
Dietary Supplement: Probiotic Clostridium butyricum CBM588® — This group received probiotic Clostridium butyricum CBM588® treatment for IBS-D as three tablets daily for 8 weeks.
  Arms: Probiotic group
Other: Standard of care IBS-D treatment — Patients in this group received standard of care IBS-D treatment of Trimebutine maleate maleate and followed a lactose-free, no-slag diet.
  Arms: Control group

SUMMARY:
Irritable bowel syndrome (IBS) is a prevalent gastrointestinal disorder affecting 15-20% of people in industrialized countries, often presenting as abdominal discomfort, pain, and altered bowel habits, significantly impacting quality of life. Among IBS subtypes, IBS-D (diarrhea-predominant) is marked by frequent, loose bowel movements, identified using the Bristol Stool Form Scale (BSFS) and classified according to Rome IV criteria. Emerging research indicates that alterations in gut microbiota, particularly a decline in butyrate-producing bacteria like *Clostridium butyricum*, play a critical role in IBS-D. Butyrate is an essential short-chain fatty acid that provides energy to colonocytes and supports intestinal health, but its deficiency may contribute to intestinal inflammation, impaired sodium and water absorption, and diarrhea. *Clostridium butyricum CBM588®* is a unique butyrate-producing bacterium that withstands oxygen, making it viable for therapeutic use. Originating from Japan, CBM588® has shown promise in enhancing gut microbiota balance, improving symptoms in IBS-D, and supporting intestinal integrity. Although primarily studied in Asian populations, additional research in Caucasian patients is warranted to validate its broader applicability and potential benefits in IBS-D symptom management.

DETAILED DESCRIPTION:
The aim of this prospective, open-label, interventional study, based on clinical data collected from real-world clinical settings, is to assess the safety and efficacy of Clostridium butyricum CBM588® in patients with IBS-D. The study consists of two cohort groups:

A cohort, where patients will receive probiotic Butirrisan® (Clostridium butyricum CBM588®) as three tablets daily, taken in the morning either before or after breakfast, for a continuous period of eight weeks.

A control cohort, consisting of IBS-D patients who received the standard of care treatment (Trimebutin maleate followed by Lactose-free, no-slag diet).

The study evaluates changes in IBS symptom severity, fecal consistency, daily frequency of evacuation and diarrhea episodes, and quality of life at the end of the treatment. The primary outcome measures include changes in the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS), fecal consistency assessed through the Bristol Stool Form Scale (BSFS), and the frequency of evacuation and diarrhea episodes. Additionally, safety will be evaluated by assessing the number of patients reporting adverse effects. The secondary outcome measure is an evaluation of quality of life, assessed using a qualitative questionnaire. Comparative analyses will be performed between the prospective Butirrisan®-treated group and the control group (Trimebutin maleate + Lactose-free, no-slag diet) to determine the relative effectiveness of probiotic therapy versus standard care.

ELIGIBILITY:
Inclusion Criteria:

* male and female, aged ≥18 years
* diagnosed with IBS-D according to the Rome IV criteria

Exclusion Criteria:

* the use of antibiotic therapies
* use of laxative therapies
* the presence of organic gastrointestinal diseases
* resection of the digestive system
* the state of pregnancy or breastfeeding
* history of drug use and alcohol abuse
* the presence of an ascertained food allergy
* the presence of lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in Irritable Bowel Syndrome Symptom Severity Scale | 8-weeks
  The scale ranges from 0 to 500, with higher scores indicating worse symptom severity. Scores are categorized as follows: 0-75 (remission), 75-174 (mild), 175-299 (moderate), and 300-500 (severe)
Changes in Fecal Consistency as assessed through the Bristol Stool Form Scale | 8-weeks
  Fecal consistency will be assessed using the Bristol Stool Form Scale, which categorizes stool from Type 1 (hard lumps) to Type 7 (liquid). Changes toward Types 3-4 indicate improvement, while shifts to Types 1 or 7 suggest worsening.
Changes in patients daily frequency of evacuation and diarrhea episodes | 8-weeks
  Probiotic effect on patients frequency of evacuation and diarrhea episodes
Number of patients reporting side effects | 8-weeks
  Safety evaluation of probiotic

SECONDARY OUTCOMES:
Changes in Quality of Life Assessment Questionnaire Score | 8-weeks
  Quality of life will be assessed through a qualitative scale with scores range from 1 to 5, with responses as follows: 1 = Not at all, 2 = Slightly, 3 = Moderately, 4 = Quite a lot, and 5 = Absolutely yes. Higher scores indicate a significant IBS impact on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Quisisana Clinic, Itala, Italy